CLINICAL TRIAL: NCT07333521
Title: Assessment of Body Composition in Children Treated With Growth Hormone for the Indication of Isolated Non-acquired Growth Hormone Deficiency.
Acronym: COMPOGHD
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP251216; 2025-A01871-48 (Other: ID RCB number)
Record Dates: First submitted 2025-12-17; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Isolated Non-acquired Growth Hormone Deficiency
Keywords: Isolated non-acquired growth hormone deficiency; Daily growth hormone therapy; Long-acting growth hormone treatments; Body mass index; Auxological measurements; Impedancemetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with isolated non-acquired growth hormone deficiency: All children in the Department of Pediatric Endocrinology, Gynecology and Diabetology at Necker Enfants Malades University Hospital treated with growth hormone, with the daily form or the delayed form, for the indication of isolated non-acquired growth hormone deficiency, naive to growth hormone treatment.
  Interventions: Other: Auxological measurements and impedancemetry

INTERVENTIONS:
Other: Auxological measurements and impedancemetry — Auxological measurements and with the Zmetric impedance meter will be carried out at each visit of the child's usual follow-up, from the day of the start of growth hormone treatment, for 3 years.

SUMMARY:
Since 1985, growth hormone deficiency (GHD) in children has been the first condition treated with daily injections of recombinant human growth hormone. Noncompliance with daily growth hormone (GH) therapy is common. Several long-acting growth hormone (LAGH) treatments have recently become available for prescription in France after pivotal phase III trials demonstrated the non-inferiority of these LAGH compared to daily GH administration. To date, published data on LAGH in children are largely limited to clinical trials of GH deficiency (GHD).

Contrary to what is observed with daily GH, body mass index increases during the first year of LAGH treatment. With the Somapacitan, the observed mean body mass index (BMI) (SDS) remained within the normal range, but with an increase from -0.17 to +0.39 in the LAGH group and a decrease from -0.25 to -0.49 in the daily GH group. In the Somatrogon study, BMI increased from -0.51 to -0.08 in the somatrogon group, while it decreased from -0.44 to -0.64 in the daily GH group. This increase in BMI was transient and then normalized over the 3-year follow-up.

In June 2025, recent data from the experience of private endocrinologists in France (AFPEL) on the real-life use of somatrogon were presented at the congress of the French Society of Pediatric Endocrinology and Diabetology. They reported a +1 SD increase in BMI during the first months of treatment in a cohort of 99 children, but an improvement was observed after prolonged treatment.

However, significant and persistent weight gain was observed in some patients, with a marked increase in abdominal adiposity. Some discontinued LAGH treatment in favor of daily GH.

Longer-term, real-life data are therefore needed to better understand the changes in BMI in these children treated with LAGH.

DETAILED DESCRIPTION:
Since 1985, growth hormone deficiency (GHD) in children has been the first condition treated with daily injections of recombinant human growth hormone. Noncompliance with daily growth hormone (GH) therapy is common. Several long-acting growth hormone (LAGH) treatments have recently become available for prescription in France after pivotal phase III trials demonstrated the non-inferiority of these LAGH compared to daily GH administration. To date, published data on LAGH in children are largely limited to clinical trials of GH deficiency (GHD).

Contrary to what is observed with daily GH, body mass index increases during the first year of LAGH treatment. With the Somapacitan, the observed mean body mass index (BMI) (SDS) remained within the normal range, but with an increase from -0.17 to +0.39 in the LAGH group and a decrease from -0.25 to -0.49 in the daily GH group. In the Somatrogon study, BMI increased from -0.51 to -0.08 in the somatrogon group, while it decreased from -0.44 to -0.64 in the daily GH group. This increase in BMI was transient and then normalized over the 3-year follow-up.

In June 2025, recent data from the experience of private endocrinologists in France (AFPEL) on the real-life use of somatrogon were presented at the congress of the French Society of Pediatric Endocrinology and Diabetology. They reported a +1 SD increase in BMI during the first months of treatment in a cohort of 99 children, but an improvement was observed after prolonged treatment.

However, significant and persistent weight gain was observed in some patients, with a marked increase in abdominal adiposity. Some discontinued LAGH treatment in favor of daily GH.

Longer-term, real-life data are therefore needed to better understand the changes in BMI in these children treated with LAGH.

The study concerns all children in the Department of Pediatric Endocrinology, Gynecology and Diabetology at Necker Enfants Malades University Hospital treated with growth hormone, with the daily form or the delayed form, for the indication of isolated non-acquired growth hormone deficiency, naive to growth hormone treatment. Auxological measurements and with the Zmetric impedance meter will be carried out at each visit of the child's usual follow-up, from the day of the start of growth hormone treatment, for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3 to 17 years inclusive.
* Confirmed diagnosis of growth hormone deficiency.
* Indication for treatment with daily or depot growth hormone.
* Growth hormone treatment naïve.- Holders of parental authority and children or adolescents informed and consenting to participate in the study.

Exclusion Criteria:

* BMI greater than +3 SD.
* Multiple pituitary insufficiency.
* Acquired growth hormone insufficiency.
* Patient with type 1 or type 2 diabetes.
* Known eating disorders.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children in the Department of Pediatric Endocrinology, Gynecology and Diabetology at Necker Enfants Malades University Hospital treated with growth hormone, with the daily form or the delayed form, for the indication of isolated non-acquired growth hormone deficiency, naive to growth hormone treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Body mass index | At the start of treatment, 3 months later, at 6 months, 12 months, 18, 24, 30 and 36 months
  Body mass index calculation at each visit of the child's usual follow-up, from the day of the start of growth hormone treatment during 3 years.

SECONDARY OUTCOMES:
Amount of muscle mass | At the start of treatment, 3 months later, at 6 months, 12 months, 18, 24, 30 and 36 months
  Description of the body composition of children treated with GH for the indication of isolated growth hormone deficiency before the start of treatment and during 3 years.
  Amount of muscle mass in kg, in %, in kg/m2.
Amount of fat mass | At the start of treatment, 3 months later, at 6 months, 12 months, 18, 24, 30 and 36 months
  Description of the body composition of children treated with GH for the indication of isolated growth hormone deficiency before the start of treatment and during 3 years.
  Amount of fat mass in kg, in %, in kg/m2.
Bone mineral content | At the start of treatment, 3 months later, at 6 months, 12 months, 18, 24, 30 and 36 months
  Description of the body composition of children treated with GH for the indication of isolated growth hormone deficiency before the start of treatment and during 3 years.
  Bone mineral content in %.
Amount of extracellular and intracellular water | At the start of treatment, 3 months later, at 6 months, 12 months, 18, 24, 30 and 36 months
  Description of the body composition of children treated with GH for the indication of isolated growth hormone deficiency before the start of treatment and during 3 years.
  Amount of extracellular and intracellular water (in L).
Hydration of fat-free mass | At the start of treatment, 3 months later, at 6 months, 12 months, 18, 24, 30 and 36 months
  Description of the body composition of children treated with GH for the indication of isolated growth hormone deficiency before the start of treatment and during 3 years.
  Hydration of fat-free mass (in %).
Description of the efficacy and tolerance of growth hormone treatment | At the start of treatment, 3 months later, at 6 months, 12 months, 18, 24, 30 and 36 months
  Description and evolution of health parameters from the patient's usual care during 3 years :
  * Weight, height, waist circumference if over 6 years old, growth rate. Tanner stage.
  * Blood pressure.
  * Clinical examination: abnormalities at injection sites, stretch marks, thyroid palpation.
  * Questionnaire on treatment tolerance: possible adverse events.
  * IGF-1 levels in ng/ml.
  * IGF-BP3 levels if available (not routinely measured).
  * Fasting blood glucose, HbA1c.
  * TSH, FT4 if available.
  * Gonadotropin, testosterone/estradiol levels if available.
  * Lipid profile : investigation of lipid abnormalities, if available.
  * Liver function tests: AST, ALT, Gamma-GT, bilirubin.

CONTACTS AND LOCATIONS:
Overall Officials: Michel MD, PhD POLAK, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Dinane MD SAMARA-BOUSTANI, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kopchick JJ, Berryman DE, Puri V, Lee KY, Jorgensen JOL. The effects of growth hormone on adipose tissue: old observations, new mechanisms. Nat Rev Endocrinol. 2020 Mar;16(3):135-146. doi: 10.1038/s41574-019-0280-9. Epub 2019 Nov 28. PMID 31780780
- [Background] de Fries Jensen L, Antavalis V, Odgaard-Jensen J, Rossi A, Pietropoli A, Hojby M. Efficacy and Safety of Somapacitan Relative to Somatrogon and Lonapegsomatropin in Pediatric Growth Hormone Deficiency: Systematic Literature Review and Network Meta-analysis. Adv Ther. 2024 Nov;41(11):4098-4124. doi: 10.1007/s12325-024-02966-y. Epub 2024 Sep 11. PMID 39261416